CLINICAL TRIAL: NCT03851224
Title: Immediate Implant Placement in Maxillary Esthetic Zone Without Augmenting the Jumping Gap Versus the Use of Autogenous Bone Particulates or Demineralized Bovine Bone Graft (Randomized Clinical Trial)
Brief Title: Immediate Implant With no Graft , Autogenous Graft or Xenograft.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa attiea, B.D.S., principal investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: immediate implants
Record Dates: First submitted 2018-09-11; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Immediate implant placement in maxillary esthetic zone without augmenting the jumping gap versus the use of autogenous bone particulates or demineralized bovine bone graft.
Who Masked: Participant
Masking Description: Immediate implant placement in maxillary esthetic zone without augmenting the jumping gap versus the use of autogenous bone particulates or demineralized bovine bone graft.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): under local anaesthesia patients hopeless teeth are be extracted. then immediate implant is palced with no graft and immediate temporary prothesis is loaded upon the immediate implants.implant stability is evaluated immediately and 3 months post operatively
  Interventions: Procedure: control group
- study group (Active Comparator): under local anaesthesia patients hopeless teeth are be extracted. then immediate implant is palced with autogenous bone graft and immediate temporary prothesis is loaded upon the immediate implants.implant stability is evaluated immediately and 3 months post operatively
  Interventions: Procedure: study group
- study group 2 (Active Comparator): under local anaesthesia patients hopeless teeth are be extracted. then immediate implant is palced withxenograft and immediate temporary prothesis is loaded upon the immediate implants.implant stability is evaluated immediately and 3 months post operatively
  Interventions: Procedure: study group 2

INTERVENTIONS:
Procedure: control group — immediate implant with immediate loading using no graft
  Arms: control group
Procedure: study group — immediate implant with immediate loading using autogenous bone graft
  Arms: study group
Procedure: study group 2 — immediate implant with immediate loading using (Geistlich Bio-Oss®) xenograft
  Arms: study group 2

SUMMARY:
Immediate implant placement with no graft , autogenous graft or xenograft with provisionalization.

DETAILED DESCRIPTION:
Immediate implant placement in maxillary esthetic zone without augmenting the jumping gap versus the use of autogenous bone particulates or demineralized bovine bone graft (Randomized Clinical Trial)

ELIGIBILITY:
Inclusion Criteria:

* patients with non-restorable teeth

Exclusion Criteria:

* intra oral pathology and systemic conditions that contraindicate dental implants.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
evaliuation of labial bone changes | 6 month
  Evaluation the thickness of the facial bony wall by millimeter in the CBCT
evaluation of marginal bone changes | 6 months
  evaluation of interproximal bone changes by millimeter in the CBCT

SECONDARY OUTCOMES:
pink aesthetic score | 6 month
  evaluation of soft tissue changes surround implant by pink aesthetic score

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M Attiea, B.S.D, Principal Investigator — Egypt Faculty of dentistry Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Al- Manial Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
web sites and papers

REFERENCES:
- [Background] Papaspyridakos P, Chen CJ, Singh M, Weber HP, Gallucci GO. Success criteria in implant dentistry: a systematic review. J Dent Res. 2012 Mar;91(3):242-8. doi: 10.1177/0022034511431252. Epub 2011 Dec 8. PMID 22157097
- [Background] Schulte W, Kleineikenscheidt H, Lindner K, Schareyka R. [The Tubingen immediate implant in clinical studies]. Dtsch Zahnarztl Z. 1978 May;33(5):348-59. German. PMID 348452
- [Background] Chen ST, Wilson TG Jr, Hammerle CH. Immediate or early placement of implants following tooth extraction: review of biologic basis, clinical procedures, and outcomes. Int J Oral Maxillofac Implants. 2004;19 Suppl:12-25. PMID 15635942
- [Background] Elian N, Cho SC, Froum S, Smith RB, Tarnow DP. A simplified socket classification and repair technique. Pract Proced Aesthet Dent. 2007 Mar;19(2):99-104; quiz 106. PMID 17491484
- [Background] Becker W, Becker BE. Guided tissue regeneration for implants placed into extraction sockets and for implant dehiscences: surgical techniques and case report. Int J Periodontics Restorative Dent. 1990;10(5):376-91. No abstract available. PMID 2098360
- [Background] Tan-Chu JH, Tuminelli FJ, Kurtz KS, Tarnow DP. Analysis of buccolingual dimensional changes of the extraction socket using the "ice cream cone" flapless grafting technique. Int J Periodontics Restorative Dent. 2014 May-Jun;34(3):399-403. doi: 10.11607/prd.1605. PMID 24804291
- [Background] Conrad EU, Gretch DR, Obermeyer KR, Moogk MS, Sayers M, Wilson JJ, Strong DM. Transmission of the hepatitis-C virus by tissue transplantation. J Bone Joint Surg Am. 1995 Feb;77(2):214-24. doi: 10.2106/00004623-199502000-00007. PMID 7844127
- [Background] Tarnow DP, Chu SJ, Salama MA, Stappert CF, Salama H, Garber DA, Sarnachiaro GO, Sarnachiaro E, Gotta SL, Saito H. Flapless postextraction socket implant placement in the esthetic zone: part 1. The effect of bone grafting and/or provisional restoration on facial-palatal ridge dimensional change-a retrospective cohort study. Int J Periodontics Restorative Dent. 2014 May-Jun;34(3):323-31. doi: 10.11607/prd.1821. PMID 24804283
- [Background] Kan JY, Rungcharassaeng K, Lozada JL, Zimmerman G. Facial gingival tissue stability following immediate placement and provisionalization of maxillary anterior single implants: a 2- to 8-year follow-up. Int J Oral Maxillofac Implants. 2011 Jan-Feb;26(1):179-87. PMID 21365054
- [Background] Chu SJ, Hochman MN, Tan-Chu JH, Mieleszko AJ, Tarnow DP. A novel prosthetic device and method for guided tissue preservation of immediate postextraction socket implants. Int J Periodontics Restorative Dent. 2014;34 Suppl 3:s9-17. doi: 10.11607/prd.1749. PMID 24956098
- [Background] Ritter AV. Xerostomia (dry mouth). J Esthet Restor Dent. 2006;18(5):306. doi: 10.1111/j.1708-8240.2006.00041.x. No abstract available. PMID 16987328
- [Background] Kan JY, Rungcharassaeng K, Lozada J. Immediate placement and provisionalization of maxillary anterior single implants: 1-year prospective study. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):31-9. PMID 12608666